CLINICAL TRIAL: NCT07313722
Title: A Randomized, Double-blind, Placebo-controlled, Dose-escalation, Single-center Phase I Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of 0.5%, 1.0%, and 1.5% BT01001 Ophthalmic Solution in Healthy Adult Volunteers
Brief Title: Study Evaluating Safety of BT01001 Ophthalmic Solution
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beyang Therapeutics Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BT01001-101
Record Dates: First submitted 2025-11-19; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- BT01001 Ophthalmic Solution dose 1 SAD (Experimental): • BT01001 Ophthalmic Solution 5 mg/ml (0.5%） N = 6 Single Ascending Dose (SAD, Day 1): 2 drops administered once to the right eye. Elution/Washout Phase: 1 day following SAD.
  Interventions: Drug: BT01001 5 mg/ml（0.5%）
- Placebo dose 1 SAD (Placebo Comparator): • Placebo Ophthalmic Solution (0 mg/mL) N = 2 Single Ascending Dose (SAD, Day 1): 2 drops administered once to the right eye. Elution/Washout Phase: 1 day following SAD.
  Interventions: Drug: Placebo
- BT01001 Ophthalmic Solution dose 1 MAD (Experimental): • BT01001 Ophthalmic Solution 5 mg/ml (0.5%） N = 6 Multiple Ascending Dose (MAD, Days 3-9): 2 drops administered twice daily (BID) from Days 3 to 8; on Day 9, 2 drops administered once in the morning only. Dose Administration: 2 drops with three minutes interval per dosing time.
  Interventions: Drug: BT01001 5 mg/ml（0.5%）
- Placebo dose 1 MAD (Placebo Comparator): • Placebo Ophthalmic Solution (0 mg/mL) N = 2 Multiple Ascending Dose (MAD, Days 3-9): 2 drops administered twice daily (BID) from Days 3 to 8; on Day 9, 2 drops administered once in the morning only. Dose Administration: 2 drops with three minutes interval per dosing time.
  Interventions: Drug: BT01001 15 mg/ml（1.5%）
- BT01001 Ophthalmic Solution dose 2 SAD (Experimental): • BT01001 Ophthalmic Solution 10 mg/ml (1.0%） N = 6 Single Ascending Dose (SAD, Day 1): 2 drops administered once to the right eye.
  Elution/Washout Phase: 1 day following SAD.
  Interventions: Drug: BT01001 10 mg/ml（1.0%）
- Placebo dose 2 SAD (Placebo Comparator): • Placebo Ophthalmic Solution (0 mg/mL) N = 2 Single Ascending Dose (SAD, Day 1): 2 drops administered once to the right eye. Elution/Washout Phase: 1 day following SAD.
  Interventions: Drug: Placebo
- BT01001 Ophthalmic Solution dose 2 MAD (Experimental): • BT01001 Ophthalmic Solution 10 mg/ml (1.0%） N = 6 Multiple Ascending Dose (MAD, Days 3-9): 2 drops administered twice daily (BID) from Days 3 to 8; on Day 9, 2 drops administered once in the morning only. Dose Administration: 2 drops with three minutes interval per dosing time.
  Interventions: Drug: BT01001 10 mg/ml（1.0%）
- Placebo dose 2 MAD (Placebo Comparator): • Placebo Ophthalmic Solution (0 mg/mL) N = 2 Multiple Ascending Dose (MAD, Days 3-9): 2 drops administered twice daily (BID) from Days 3 to 8; on Day 9, 2 drops administered once in the morning only. Dose Administration: 2 drops with three minutes interval per dosing time.
  Interventions: Drug: Placebo
- BT01001 Ophthalmic Solution dose 3 SAD (Experimental): • BT01001 Ophthalmic Solution 15 mg/ml (1.5%） N = 6 Single Ascending Dose (SAD, Day 1): 2 drops administered once to the right eye.
  Elution/Washout Phase: 1 day following SAD.
  Interventions: Drug: BT01001 15 mg/ml（1.5%）
- Placebo dose 3 SAD (Placebo Comparator): • Placebo Ophthalmic Solution (0 mg/mL) N = 2 Single Ascending Dose (SAD, Day 1): 2 drops administered once to the right eye. Elution/Washout Phase: 1 day following SAD.
  Interventions: Drug: Placebo
- BT01001 Ophthalmic Solution dose 3 MAD (Experimental): • BT01001 Ophthalmic Solution 15 mg/ml (1.5%） N = 6 Multiple Ascending Dose (MAD, Days 3-9): 2 drops administered twice daily (BID) from Days 3 to 8; on Day 9, 2 drops administered once in the morning only. Dose Administration: 2 drops with three minutes interval per dosing time.
  Interventions: Drug: BT01001 15 mg/ml（1.5%）
- Placebo dose 3 MAD (Placebo Comparator): • Placebo Ophthalmic Solution (0 mg/mL) N = 2 Multiple Ascending Dose (MAD, Days 3-9): 2 drops administered twice daily (BID) from Days 3 to 8; on Day 9, 2 drops administered once in the morning only. Dose Administration: 2 drops with three minutes interval per dosing time.
  Interventions: Drug: Placebo
- BT01001 Ophthalmic Solution dose 4 MAD (Experimental): • BT01001 Ophthalmic Solution 15 mg/ml (1.5%） N = 6 Multiple Ascending Dose (MAD, Days 1-7): 2 drops administered three times daily (TID) from Days 1 to 6; on Day 7, 2 drops administered once in the morning only to the right eye.
  Dose Administration: 2 drops with three minutes interval per dosing time.
  Interventions: Drug: BT01001 15 mg/ml（1.5%）
- Placebo dose 4 MAD (Placebo Comparator): • Placebo Ophthalmic Solution (0 mg/mL) N = 2 Multiple Ascending Dose (MAD, Days 1-7): 2 drops administered three times daily (TID) from Days 1 to 6; on Day 7, 2 drops administered once in the morning only to the right eye.
  Dose Administration: 2 drops with three minutes interval per dosing time.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BT01001 5 mg/ml（0.5%） — BT01001 Ophthalmic Solution will be administered as topical instillation into the right eye of each subject according to the assigned dosing schedule.
  Other Names: BT01001 Ophthalmic Solution
  Arms: BT01001 Ophthalmic Solution dose 1 MAD; BT01001 Ophthalmic Solution dose 1 SAD
Drug: BT01001 10 mg/ml（1.0%） — BT01001 Ophthalmic Solution will be administered as topical instillation into the right eye of each subject according to the assigned dosing schedule.
  Other Names: BT01001 Ophthalmic Solution
  Arms: BT01001 Ophthalmic Solution dose 2 MAD; BT01001 Ophthalmic Solution dose 2 SAD
Drug: BT01001 15 mg/ml（1.5%） — BT01001 Ophthalmic Solution will be administered as topical instillation into the right eye of each subject according to the assigned dosing schedule.
  Other Names: BT01001 Ophthalmic Solution
  Arms: BT01001 Ophthalmic Solution dose 3 MAD; BT01001 Ophthalmic Solution dose 3 SAD; BT01001 Ophthalmic Solution dose 4 MAD; Placebo dose 1 MAD
Drug: Placebo — Placebo BT01001 Ophthalmic Solution will be administered as a topical instillation into the right eye of each subject following the same dosing schedule as the active treatment.
  Other Names: BT01001 Ophthalmic Solution Placebo
  Arms: Placebo dose 1 SAD; Placebo dose 2 MAD; Placebo dose 2 SAD; Placebo dose 3 MAD; Placebo dose 3 SAD; Placebo dose 4 MAD

SUMMARY:
This Phase I study is designed to evaluate the safety, tolerability, and pharmacokinetic profile of BT01001 Ophthalmic Solution in healthy adult volunteers. The primary objectives are to assess the safety and tolerability of single and multiple ascending doses and to characterize the pharmacokinetics of BT01001 Ophthalmic Solution following topical ocular administration.

This is a randomized, double-blind, placebo-controlled, dose-escalation trial consisting of four ascending dose cohorts. Each cohort will enroll eight participants, including six receiving BT01001 Ophthalmic Solution and 2 receiving Placebo.

ELIGIBILITY:
Inclusion Criteria:

-

General Inclusion Criteria:

1. Healthy male or female participant, 18 to 50 years of age at the time of screening, who are in good health based on medical history, physical examinations, vital signs, electrocardiogram (ECG), and clinical laboratory evaluations.
2. Body Mass Index (BMI) between 18.0 and 27.0 kg/m² (inclusive).
3. Negative alcohol breath test and negative urine drug screen at screening.
4. Willing and able to comply with all study procedure and capable of good communication with study personnel.
5. Participants of childbearing potential must agree to abstain from sexual intercourse or use an effective method of contraception from screening until 90 days after the final study drug administration; Female participants of childbearing potential must have a negative urine pregnancy test at screening.
6. Able to understand the study procedure and voluntarily sign the written informed consent form.

   Ophthalmology Inclusion Criteria:
7. Corrected vision acuity ≥ 0.8 in both eyes.
8. Intraocular pressure (IOP) < 21 mmHg in each eye, with and inter-eye difference < 4 mmHg.
9. Slit-lamp and ophthalmoscopic examinations that are normal or show abnormalities considered not clinically significant by the investigator.

Exclusion Criteria:

-

General Exclusion Criteria:

1. Known or suspected hypersensitivity to any component of the investigational product, or a history of multiple allergies two or more allergens).
2. History or presence of any clinically significant diseases or abnormality, including but not limited to cardiovascular, cerebrovascular, respiratory, endocrine, metabolic, renal, hepatic, gastrointestinal, dermatologic, oncologic, hematologic, immunologic, infectious, neurologic or psychiatric conditions, or any acute or chronic condition that may interfere with study assessments.
3. Participation in any investigational drug or medical device trial within 90 days prior to study drug administration.
4. Use of prescription or over-the-counter medications within 14 days prior to dosing, or unwillingness to discontinue such medications during the study.
5. Receipt of systemic corticosteroid therapy within 6 months prior to dosing.
6. History of alcohol abuse or substance abuse within 2 years prior to dosing.
7. Regular smoking of ≥ 5 cigarettes per day (or equivalent tobacco use) within 12 weeks prior to screening, or inability/unwillingness to abstain during the study.
8. Average alcohol consumption >14 units per week within 12 weeks prior to screening (1 unit approximately equivalent to 360 mL beer, 150 mL wine, or 45 mL of 40% spirits).
9. History or evidence of intravenous illicit drug use; positive test for HIV, HCV, HBsAg, anti-HCV, anti-HIV, or Treponema pallidum antibody at screening.
10. Blood donation or receipt of blood products within 30 days prior to dosing.
11. History of bleeding disorders or coagulation abnormalities.
12. Clinically significant abnormalities on physical examination, vital signs, 12-lead ECG, or laboratory results at screening.

    Abnormal findings that normalize on repeat testing may be accepted if assessed not clinically significant by the investigator.
13. Current or past use of bariatric medications or history of bariatric surgery (e.g., gastric bypass).
14. Impaired mental status or other factors that may compromise adherence to study requirements.
15. Any conditions that, in the investigator's judgment, may interfere with study assessments or pose the participant to unacceptable risks.

    Ophthalmology Exclusion Criteria:
16. History of ocular surgery, ocular trauma, or chronic eye disease.
17. Current use of contact lenses or use within 2 weeks prior to first dosing.
18. Ocular abnormalities or symptoms considered clinically significant by the investigator.
19. Use of intraocular injectable or implantable therapies, or topical ophthalmic medications, within 2 months prior to dosing, or expected need during the study.
20. History or evidence of ocular e infection, inflammation, blepharitis, or conjunctivitis within 2 months; history of herpes simplex keratitis.
21. Clinically significant findings on ophthalmic evaluations (slit lamp, BCVA, IOP, OCT/OCTA, or fundus examination) that, in the investigator's judgment, may interfere with ocular safety evaluations.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events as Assessed by CTCAE V5.0 | after dosing up to 14 days/12 days
  Any AE event related to study treatment
Dose-Limiting Toxicity | SAD: after dosing up to 2 days; MAD: after dosing up to 8 days
  ≥CTCAE 2 ocular adverse events or· >CTCAE 3 non-ocular· adverse events· assessed with·CTCAE·5.0

SECONDARY OUTCOMES:
Measured Area Under the Curve (AUC) | SAD(dose 1-3): Day 1, Day 2; MAD(dose 1-3): Day 8, Day 9, Day 10; MAD(dose 4): Day 6, Day 7,Day 8;
  SAD(dose 1-3): at Day 1 pre-dose, 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 24h.
  MAD(dose 1-3): at Day 8 pre-dose(before the first dose), Day 8 pre-dose(before the second dose), Day 9 pre-dose(before the first drop), 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 24h.
  MAD(dose 4): at Day 6 pre-dose(before the second dose), Day 6 pre-dose(before the third dose), Day 7 pre-dose(before the first dose), 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 24h.
Time to Maximum Plasma Concentration (Tmax) | SAD(dose 1-3): Day 1, Day 2; MAD(dose 1-3): Day 8, Day 9, Day 10; MAD(dose 4): Day 6, Day 7,Day 8;
  SAD(dose 1-3): at Day 1 pre-dose, 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 24h.
  MAD(dose 1-3): at Day 8 pre-dose(before the first dose), Day 8 pre-dose(before the second dose), Day 9 pre-dose(before the first drop), 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 24h.
  MAD(dose 4): at Day 6 pre-dose(before the second dose), Day 6 pre-dose(before the third dose), Day 7 pre-dose(before the first dose), 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 24h.
Maximum Plasma Concentration (Cmax) | SAD(dose 1-3): Day 1, Day 2; MAD(dose 1-3): Day 8, Day 9, Day 10; MAD(dose 4): Day 6, Day 7,Day 8;
  SAD(dose 1-3): at Day 1 pre-dose, 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 24h.
  MAD(dose 1-3): at Day 8 pre-dose(before the first dose), Day 8 pre-dose(before the second dose), Day 9 pre-dose(before the first drop), 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 24h.
  MAD(dose 4): at Day 6 pre-dose(before the second dose), Day 6 pre-dose(before the third dose), Day 7 pre-dose(before the first dose), 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 24h.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, China